CLINICAL TRIAL: NCT01956487
Title: A Phase 1, Open-Label, Crossover Study to Demonstrate the Bioequivalence of RYTHMOL SR® (Propafenone Hydrochloride) Manufactured at Two Different Sites
Brief Title: Bioequivalence of RYTHMOL SR® Manufactured at Two Different Sites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 116371
Record Dates: First submitted 2012-07-19; First posted 2013-10-08 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Arrhythmia, Cardiac
Keywords: Bioequivalence; RYTHMOL SR®; Atrial fibrillation; Propafenone; Pharmavokinetics
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Propafenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propafenone (Other): Open label comparison of 2 formulations
  Interventions: Drug: Propafenone

INTERVENTIONS:
Drug: Propafenone — Comparison of drug from 2 manufacturing sites

SUMMARY:
Bioequivalence of propafenone hydrochloride capsules manufactured at two different sites

DETAILED DESCRIPTION:
This will be a Phase 1, randomized, open-label, single-dose, three-period, crossover study to assess the bioequivalence of propafenone hydrochloride manufactured at two different sites in healthy adult volunteers. Approximately 36 subjects will receive a 3 single doses of propafenone hydrochloride 425mg, each administered separately, in the fasted state with a 7 day washout period between doses. Propafenone hydrochloride is an antiarrhythmic indicated to prolong the time to recurrence of symptomatic atrial fibrillation in patients with episodic (most likely paroxysmal or persistent) atrial fibrillation who do not have structural heart disease. A follow-up visit will occur 7-10 days after the final dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Body weight greater than or equal to 50kg and BMI within the range 18.5 - 31.0kg/m2 (inclusive).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* A female subject is eligible to participate if she postmenopausal or on a stable regimine of an approved contracetive
* Capable of giving written informed consent,

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12g of alcohol: 12 ounces (360ml) of beer, 5 ounces (150ml) of wine or 1.5 ounces (45ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: either 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* The subject has donated blood or blood products in excess of 500mL within a 56 day period.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Unwilling to abstain from alcohol for 48 hours prior to screening and 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* The subject's systolic blood pressure is outside the range of 90-140 mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 55-100bpm for female subjects or 50-100bpm for male subjects.
* Screening ECG within normal limts for age and gender
* Evidence of previous myocardial infarction.
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome, non-sustained or sustained ventricular tachycardia (3 or more consecutive ventricular ectopic beats), sinus pauses > 3 seconds, or other significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04-11 (Actual); Primary Completion 2012-06-27 (Actual); Study Completion 2012-06-27 (Actual)

PRIMARY OUTCOMES:
Bioequvalence | 48 hours
  Two formulations of propafenone hydrochloride

SECONDARY OUTCOMES:
Pharmacokinetics | 48 hours
  Plasma AUC and Cmax of propafenone
Adverse events | 48 hours
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] "RYTHMOL is a registered trademark of G. Petrik used under license by Abbott Laboratories."
- See also: Results for study 116371 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116371?search=study&search_terms=116371#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 116371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register